CLINICAL TRIAL: NCT07279519
Title: Predictive Value of the Clinical Frailty Scale, Katz ADL, and Admission Laboratory Markers for Postoperative ICU Mortality in Geriatric Patients: A Prospective Observational Study
Brief Title: Predictive Value of Frailty Scores and Admission Laboratory Markers for Postoperative ICU Mortality
Acronym: GERI-MORTAL
Status: Not yet recruiting | Type: Observational
Sponsor: Malatya Egitim Ve Arastirma Hastanesi (Other Government)
Responsible Party: Principal Investigator, Leman Acun Delen, Associate Professor of Anesthesiology and İntensive Care, Malatya Egitim Ve Arastirma Hastanesi
Other Study IDs: MEAH-GER-ICU-2025-01
Record Dates: First submitted 2025-11-26; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Mortality; Frailty at Older Adults; Activities of Daily Living; Postoperative Complications
Keywords: Frailty; ICU Mortality; Geriatric Surgery
MeSH Terms: conditions — Postoperative Complications; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geriatric Postoperative ICU Cohort: This cohort includes geriatric patients (≥65 years) admitted to the intensive care unit after surgery. All participants are followed prospectively to evaluate clinical frailty, functional status, and admission laboratory parameters in relation to postoperative ICU mortality.

SUMMARY:
This prospective observational study aims to evaluate the predictive value of the Clinical Frailty Scale (CFS), the Katz Activities of Daily Living (ADL) scale, and admission laboratory markers for postoperative mortality among geriatric patients admitted to the intensive care unit (ICU) after surgery. Frailty assessment and functional status are increasingly recognized as determinants of outcomes in older adults, yet their combined predictive power with routine laboratory parameters at ICU admission remains unclear. By systematically collecting clinical scores and laboratory data at the time of ICU admission, this study seeks to identify early predictors of mortality and support risk-stratification in geriatric postoperative patients.

DETAILED DESCRIPTION:
This prospective observational study aims to evaluate the predictive value of the Clinical Frailty Scale (CFS), Katz Activities of Daily Living (ADL) score, and admission laboratory markers for postoperative ICU mortality in geriatric patients. Frailty and functional dependency are known to influence postoperative outcomes; however, their combined role alongside early biochemical indicators at the time of ICU admission has not been well defined in this population.

In this study, patients aged 65 years and older who are admitted to the intensive care unit following surgery will be assessed using the CFS and Katz ADL scores within the first hours of ICU admission. Laboratory data obtained at the time of admission-including complete blood count, renal and hepatic panels, electrolytes, markers of inflammation, and arterial blood gas parameters-will be recorded. Patients will subsequently be followed throughout their ICU stay to document clinical course and outcomes, with ICU mortality designated as the primary endpoint.

The goal of this research is to identify which frailty indicators and laboratory markers are independently associated with mortality, and to explore whether combining functional status scores with early laboratory abnormalities improves risk stratification in geriatric postoperative ICU patients. The findings may support the development of simple, bedside-applicable tools for early mortality prediction and clinical decision-making in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

Individuals aged 65 years and older Undergoing elective or emergency surgery Monitored in the intensive care unit for at least 24 hours after surgery Provision of informed consent by the patient or the legal representative

Exclusion Criteria:

Patients with incomplete or unavailable data sets ICU stays shorter than 24 hours Patients admitted for organ transplantation or those in the terminal stage receiving palliative care

Ages: 65 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: This study will include geriatric patients aged 65 years and older who have undergone elective or emergency surgery and require postoperative monitoring in the intensive care unit for at least 24 hours. Patients must provide informed consent personally or through a legally authorized representative
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
30-day ICU Mortality | 30 days after ICU admission
  Mortality status will be determined at the time of ICU discharge. Mortality is defined as all-cause death occurring during the postoperative ICU stay. Data will be collected prospectively from the electronic medical record and verified by the ICU clinical team. The outcome will be recorded as a binary variable (survived / died)

SECONDARY OUTCOMES:
Rate of ICU Length of Stay in Geriatric Postoperative Patients | From ICU admission to ICU discharge (up to 28 days)
  Duration of stay in the intensive care unit, recorded in days. Longer ICU stay is often associated with increased frailty, limited functional capacity, and higher physiological burden. This variable will be extracted from the clinical records and analyzed in relation to frailty, Katz ADL score, and admission laboratory markers.
Association Between Laboratory Markers and Frailty Scores | At ICU admission
  Correlation analysis between baseline laboratory parameters (e.g., hemoglobin, creatinine, CRP, albumin) and frailty assessments (Clinical Frailty Scale and Katz ADL).

CONTACTS AND LOCATIONS:
Overall Officials: Leman Acun Delen, MD, Assoc. Prof., Principal Investigator — Malatya Training and Research Hospital, Department of Anesthesiology and Intensive Care
Locations (1):
- Malatya Eğitim Araştırma Hastanesi, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to institutional policies, patient privacy concerns, and local ethical regulations, individual-level clinical data cannot be shared publicly. Only aggregated and anonymized results will be reported.

REFERENCES:
- [Result] Csiszar A, Ungvari Z, Edwards JG, Kaminski P, Wolin MS, Koller A, Kaley G. Aging-induced phenotypic changes and oxidative stress impair coronary arteriolar function. Circ Res. 2002 Jun 14;90(11):1159-66. doi: 10.1161/01.res.0000020401.61826.ea. PMID 12065318
- [Result] Moisi L, Mino JC, Guidet B, Vallet H. Frailty assessment in critically ill older adults: a narrative review. Ann Intensive Care. 2024 Jun 18;14(1):93. doi: 10.1186/s13613-024-01315-0. PMID 38888743
- [Result] Chen W, Chen M, Qiao X. Interaction of lactate/albumin and geriatric nutritional risk index on the all-cause mortality of elderly patients with critically ill heart failure: A cohort study. Clin Cardiol. 2023 Jul;46(7):745-756. doi: 10.1002/clc.24029. Epub 2023 May 24. PMID 37226575